CLINICAL TRIAL: NCT01875328
Title: Stroke Therapy, Education, Prevention: Telemedicine Outpatient Initiative Trial
Acronym: STEP TO IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9011
Record Dates: First submitted 2013-06-06; First posted 2013-06-11 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Stroke
Keywords: stroke; blood pressure; telemedicine
MeSH Terms: conditions — Stroke | interventions — Telemedicine; Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemedicine (Experimental): Telemedicine group
  Interventions: Other: Telemedicine
- Clinic (Active Comparator): Clinic group
  Interventions: Other: Clinic

INTERVENTIONS:
Other: Telemedicine — Post stroke follow up in home using telemedicine.
  Arms: Telemedicine
Other: Clinic — Post stroke clinic group follow up
  Arms: Clinic

SUMMARY:
This study aims to determine whether patients who have had a stroke caused by a blockage of blood flow to the brain can have medical follow up after they leave the hospital in their home using a camera connected to a computer, also called telemedicine. Patients who have follow-up with telemedicine will be compared with patients following up in the usual way, by coming to clinic, and will have the same expectations for medical care and lifestyle changes like quitting smoking, exercising, and controlling their cholesterol. The study will try to show those stroke patients who live 75 miles or more from Oregon Health & Science University (OHSU) and use a computer for follow up: 1) Will be able to complete the recommended visits using telemedicine in the home as well as those who come to clinic; 2) Will have blood pressures controlled at one year's time as well as those who follow up in the usual way by coming into clinic; 3) The patients followed with telemedicine will be as satisfied with the type of follow up they had as those followed in the usual way in the clinic. In the future, more patients who live at a distance from a major hospital might be able to get quality stroke care follow up using telemedicine if the study finds that telemedicine does meet these goals.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 and over.
2. Diagnosis of ischemic stroke or transient ischemic attack (TIA).
3. mRS≤3 or discharged home or inpatient rehabilitation with the intention to return home with reliable caregiver, regardless of mRS score.
4. Patient is willing and able to comply with all follow up visits for the protocol.
5. Patient available by phone.
6. Patient or caregiver must be able to operate an automated blood pressure cuff.
7. Patients living beyond a 75 mile radius must have private access to a computer to facilitate in-home telemedicine follow up visits.

Exclusion Criteria:

1. History of uncontrolled severe hypertension or refractory to medical management.
2. Severe liver impairment (AST or ALT > 3x normal).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Outpatient stroke follow-up after discharge using telemedicine in the home is feasible as assessed by visit and intervention adherence for patients living outside a 75 mile radius from OHSU. | up to 1 year

SECONDARY OUTCOMES:
Patients being followed in the telemedicine group will achieve rates of goal blood pressure similar to those being followed in clinic. | 30 days, 1 year

OTHER OUTCOMES:
Patients being followed in the telemedicine group will have similar rates of satisfaction with the follow up regimen compared to those in the traditional clinic follow up group. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Darren Larsen, RN, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States